CLINICAL TRIAL: NCT01094210
Title: Evaluation of a Low-fluoride Anticaries Toothpaste Containing an Innovative Calcium Technology
Brief Title: Evaluation of a Low-fluoride Anticaries Toothpaste
Status: Completed | Type: Observational
Sponsor: Indiana Nanotech, LLC (Other)
Collaborators: The University of Texas Health Science Center at San Antonio (Other)
Responsible Party: Principal Investigator, Dr. Robert L. Karlinsey, Managing Member, Indiana Nanotech, LLC
Other Study IDs: 1R43DE020998-01 (NIH)
Record Dates: First submitted 2010-03-25; First posted 2010-03-26 (Estimated); Last update posted 2015-03-25 (Estimated); Status verified 2011-06

CONDITIONS: Tooth Abnormality
Keywords: Anti-erosion dental benefits
MeSH Terms: conditions — Tooth Abnormalities | interventions — Fluorides, Topical

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- G1: 500 ppm F Test Toothpaste
  Interventions: Drug: Fluorides, Topical
- G2: 1100 ppm F Control Toothpaste
  Interventions: Drug: Fluorides, Topical

INTERVENTIONS:
Drug: Fluorides, Topical — 500 ppm F and 1100 ppm F topical toothpastes comprise sodium fluoride in each.

SUMMARY:
The purpose of this trial is to evaluate the anticaries remineralizing potential of a toothpaste containing 500 ppm fluoride plus fTCP technology relative to a commercially available toothpaste via a double-blind cross-over in situ (or intra-oral) clinical model, whereby approved human participants will wear an orthodontic appliance fitted with an enamel specimen for the duration of a leg (28 days). There will be two test legs.

ELIGIBILITY:
Inclusion Criteria:

* 30 adult subjects (between 18-50 years of age)

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: This in situ study will recruit 30 adult subjects (between 18-50 years of age). No potential subject will be excluded from this study, regardless of their gender or racial/ethnic origins. However, it is expected that about 18 (60%) of the 30 subjects in the trial will be women. This distribution will allow for meaningful comparisons between gender groups. We will recruit patients attending the clinics of UTHSCSA dental school clinics, which reflect the ethnic mix of the area the clinics serve. However, majority of subjects will be Hispanic due to the high Hispanic prevalence (57.8%) in San Antonio. Thus, minorities will be included at a similar rate to that in the general population attending for dental care,
Sampling Method: Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2010-09; Primary Completion 2011-03 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
Surface Microhardness | 30 days
  Strength measurements made at the enamel surface of the enamel specimen
Transverse Microradiography | 30 days
  X-ray analysis of enamel lesion
Cross-Sectional Microhardness | 30 days
  Strength measurements made within the enamel lesion of the enamel specimen

CONTACTS AND LOCATIONS:
Locations (1):
- Dental Diagnostic Clinic within the University of Texas Health Science Center, San Antonio, Texas, United States